CLINICAL TRIAL: NCT05800340
Title: Neoadjuvant Toripalimab Combined With Chemotherapy in Rare Mutations Stage IIB-IIIB NSCLC
Brief Title: Neoadjuvant Immunotherapy in Rare Mutations Localized NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEORM
Record Dates: First submitted 2023-03-21; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Non-Small Cell Lung Cancer; RET Driver Mutation; BRAF V600 Mutation; Erb-B2 Receptor Tyrosine Kinase Exon 20 Mutation; MET Amplification; MET Exon 14 Skipping Mutation
Keywords: Non-small Cell Lung Cancer; Neoadjuvant immunotherapy; Rare Mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — toripalimab; Taxes; Pemetrexed; Carboplatin

STUDY DESIGN:
Intervention Model Description: 3 cycles of neoadjuvant Toripalimab (240mg every 3 weeks) with nab-paclitaxel + carboplatin, or pemetrexed + carboplatin (decided by investigators; nab-paclitaxel 135 mg/m2, d1, 8 and carboplatin AUC 5, d1 every 3 weeks; pemetrexed, 500mg/m2 d1 every 3 weeks) will be administered before surgery, followed by optional adjuvant treatment including chemotherapy for 3-4 cycles or rare mutations-TKIs for up to 2 year or till disease progression or unacceptable toxicity.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab plus chemotherapy (Experimental): 3 cycles of neoadjuvant Toripalimab (240mg every 3 weeks) with nab-paclitaxel + carboplatin, or pemetrexed + carboplatin (decided by investigators; nab-paclitaxel 135 mg/m2, d1, 8 and carboplatin AUC 5, d1 every 3 weeks; pemetrexed, 500mg/m2 d1 every 3 weeks) will be administered before surgery, followed by optional adjuvant treatment including chemotherapy for 3-4 cycles or rare mutations-TKIs for up to 2 years or till disease progression or unacceptable toxicity.
  Interventions: Biological: Toripalimab; Drug: Nab paclitaxel; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Biological: Toripalimab — 240mg Q3W
Drug: Nab paclitaxel — 135 mg/m2, d1, 8 Q3W
Drug: Pemetrexed — 500mg/m2, d1 Q3W
Drug: Carboplatin — AUC 5, d1 Q3W

SUMMARY:
Phase II, single-arm, open-label single center study that assess clinical feasibility and safety of 3 cycles neoadjuvant Toripalimab plus chemotherapy in rare mutations stage IIB-IIIB NSCLC followed by optional adjuvant treatment upon investigators' decisions.

DETAILED DESCRIPTION:
30 eligible patients will be enrolled and 3 cycles of Toripalimab 240mg + chemotherapy (Nab-paclitaxel + carboplatin, or pemetrexed + carboplatin) will be administered. Rare mutations include RET fusions, BRAF (V600E or non-V600E but confirmed driver mutations), ERBB2 exon20 insertion, MET amplification (FISH confirmed) or exon 14 skipping. Dynamic blood samples before, during or after neoadjuvant treatment will be obtained for exploratory analysis. Patients who showed inferior response to neoadjuvant treatment leading to unresectable disease will be scheduled for local radiation or other potential subsequent treatment regarding multidisciplinary discussion. After completion of local treatment (surgery or radiation), patients will be provided with optional adjuvant treatment including chemotherapy or/and rare mutations TKI upon investigators' consideration. The primary objective of the study is pathological complete response (pCR) defined as no residue tumor found in both primary lung cancer and metastatic lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 Years and older
2. ECOG physical score 0-1 points; expected survival time ≥ 3 months;
3. Pathologically confirmed diagnosis with Stage IIB-IIIB NSCLC which harbored rare driver alteration including RET fusions, BRAF (V600E or non-V600E but confirmed driver mutations), ERBB2 exon20 insertion, MET amplification (FISH confirmed) or exon 14 skipping. Suspected N2 disease should be confirmed by either mediastinoscopy or EBUS. N1 disease could be determined through PET/CT but biopsy of primary lung cancer is needed;
4. Lung function capacity capable of tolerating the proposed lung surgery
5. Available tissue of tumor for PD-L1 test
6. Subjects voluntarily joined the study and signed informed consent, with good compliance to follow-up.

Exclusion Criteria:

1. Stage I and stage IV NSCLC;
2. Patients who have previously used any other anti-tumor drugs or radiotherapy;
3. Large panel NGS indicated sensitive EGFR alteration, ALK fusion, ROS1 fusion or any other driver mutations combined with MDM2/MDM4 amplification;
4. Histologically confirmed small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer);
5. A history of active bleeding within the 6 months before enrollment, or receiving thrombolysis or anticoagulant therapy, or the investigator believes that there is a clear tendency to gastrointestinal bleeding (such as esophageal varices with bleeding risk, local activity) Ulcer lesions, etc.) or active hemoptysis;
6. Patients with any underlying disease that investigators consider it may affect patient's prognosis including sever cardiovascular, pulmonary disease or serious infections; Clinically obvious gastrointestinal abnormalities, which may affect the intake, transport or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or patients with total gastrectomy;
7. Known or suspected autoimmune disease with activity. Participants may be enrolled if they have type 1 diabetes, hypothyroidism that requires only hormone replacement therapy, skin diseases that require no systemic treatment (such as purpura, psoriasis, or hair loss), or other conditions that are not expected to return without external trigger.
8. Patients with active hepatitis B (positive for HBsAg) or hepatitis C (positive for HCV RNA).
9. Patients with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)
10. Patients with other active malignancies within five years
11. Pregnant or lactating women; those who have fertility are unwilling or unable to take effective contraceptive measures;
12. Patients with low compliance or willingness to take the drugs and surveillance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | pCR will be assessed within 2 weeks after surgery
  Evaluation of the pathological complete response: The pathological complete response is defined as the absence of residual tumor in both lung and lymph nodes after neoadjuvant treatment.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) | MPR will be assessed within 2 weeks after surgery
  Percentage of Participants with Major Pathologic Response. MPR was defined as percentage of tumor cells within tumor bed less than 10% for both primary lung lesions and metastatic lymph nodes.
Event-Free Survival (EFS) | From date of initiation of neoadjuvant treatment to disease progression, reoccurrence, or death due to any cause, up to 36 months.
  Event-free survival (EFS) is defined as the length of time from initiation of neoadjuvant treatment to any of the following events: any progression of disease precluding surgery, progression or recurrence disease based on response evaluation criteria in solid tumors (RECIST) 1.1 after surgery, or death due to any cause.
Overall Survival (OS) | From date of initiation of neoadjuvant treatment to the date of all-cause death, assessed up to 60 months.
  Overall survival (OS) is defined as the time between the date of initiation of neoadjuvant treatment and the date of death.
Adverse Events (AEs) | From date of initiation of neoadjuvant treatment till treatment discontinuation, assessed up to 14 weeks.
  Incidence of all grade AE which has been confirmed to be correlated with neoadjuvant treatment or surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences, Guanzhou, Guangdong, China